CLINICAL TRIAL: NCT04525911
Title: Assessment of Long-term Impact Post COVID-19 for Patients and Health Care Professionals of the European Hospital
Acronym: ALCOVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020- A01647-32
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptomatic COVID-19 infection confirmed or probable: Patients and medical staff having symptomatic COVID-19 infection confirmed (by RT-PCR or ELISA serology) or probable (CT criteria)
  Interventions: Diagnostic Test: Diagnostic Test: serology test for COVID-19

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: serology test for COVID-19 — a serology test will be performed at M3

SUMMARY:
The purpose of the study is to Assess of Long-term impact post COVID for patients and health care professionals.The patients and medical staff will be followed for 2 years in order to provide clinical and paraclinical data not yet published in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years,
* Symptomatic COVID-19 infection confirmed (by RT-PCR or ELISA serology) or probable (CT criteria),
* Having given free and informed written consent,
* Being affiliated with or benefiting from a social security scheme.
* Patients / caregivers may be included in several ancillary studies at the same time.

Exclusion Criteria:

-Subject to a measure for the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient and medical staff with confirmed or probable COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of post-traumatic stress symptoms (Post traumatic Stress Disorder (PTSD) scale) at M3 for patients and caregivers | 3 months
  measure used to assess symptoms of post-traumatic stress disorder. Individuals should rate their experience with each of the 17 symptoms of PTSD on a scale of 1 to 5 (1 = not at all, 2 = a little, 3 = moderately, 4 = a little, and 5 = extremely) versus to a specific traumatic event

SECONDARY OUTCOMES:
Evaluation of post-traumatic stress symptoms (PTSD scale) at M12 and M24 for patients and caregivers | 12 and 24 months
Change from M3 in the score of the mental (MCS), physical (PCS) components and the scores of the individual domains of the questionnaire SF36 to M12 and M24 for the entire study population | 12 and 24 months
% of patients presenting a positive result by ELISA serology (= without distinction of IgG, IgM and IgA) | 3 months
Comparison of M0 chest CT results at each follow-up for the entire study population | 24 months

OTHER OUTCOMES:
Change from M3 score measuring anxiety (HAD-A) and depression score (HAD-D) to M12 and M24 for patients and caregivers. | 12 and 24 months
  HAD-A score measuring anxiety (example "I feel tense or nervous") and HAD-D score for depression (example "I have the impression of operating in slow motion").
  * 7 or less: no symptoms
  * 8 to 10: doubtful symptomatology
  * 11 and more: definite symptomatology.
Change from M3 in the B-IPQ score at M12 and M24 for patients and caregivers. | 12 and 24 months
  The Brief Illness Perception Questionnaire (B-IPQ) includes 9 items that assess different components of "perception of the disease"( score 0 to 10 for each items)
Evaluation of the microbiotic signature according to the severity of the disease at M3, M6 and M12 | 6 and 12 months
Evaluation of the fatigue EVA score and quality of life (SF36) at M6 and M12 | 6 and 12 months
  score from 0 to 10 (0 not tired, 10 max tired)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé PEGLIASCO, Principal Investigator — Hôpital Europeen Marseille
Locations (1):
- BENNANI, Marseille, France

IPD SHARING:
Plan to Share IPD: No